CLINICAL TRIAL: NCT06381245
Title: First-time Ablation of Atrial Fibrillation Registry
Acronym: DIPE
Status: Recruiting | Type: Observational
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: KB/265/2023
Record Dates: First submitted 2024-04-18; First posted 2024-04-24 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-02

CONDITIONS: Atrial Fibrillation; Arrhythmia
Keywords: Atrial fibrillation; Arrhythmia; Pulsed field ablation; Radiofrequency ablation; Catheter ablation; Prediction; Detection; Mobile Health; Telemedicine
MeSH Terms: conditions — Atrial Fibrillation; Arrhythmias, Cardiac

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: PPG-based remote heart rhythm/rate monitoring — PPG-based remote heart rhythm/rate monitoring
Diagnostic Test: ECG-based remote heart rhythm/rate monitoring — ECG-based remote heart rhythm/rate monitoring
Diagnostic Test: Transthoracic and transesophageal echocardiography examination — Transthoracic and transesophageal echocardiography examination
Diagnostic Test: Liver ultrasound examination — Liver ultrasound examination
Diagnostic Test: Rotational angiography with three-dimensional reconstruction — Rotational angiography with three-dimensional reconstruction
Diagnostic Test: Blood-derived biomarker analysis — Blood-derived biomarker analysis
Diagnostic Test: Mobile health-based spirometry — Mobile health-based spirometry

SUMMARY:
Atrial fibrillation (AF) is a prevalent cardiac arrhythmia affecting millions globally, with projections indicating a doubling of cases by 2050. AF is linked to heightened cardiovascular risks like stroke and increased healthcare costs. Ablation, targeting the arrhythmia substrate, is a method to manage AF, yet recurrence rates remain high (20-45% in the first year). Studies highlight the impact of comorbidities, AF characteristics, ablation techniques, and myocardial remodeling markers on AF progression and ablation efficacy. However, there's no definitive guidance on selecting these factors for predicting treatment success.

The aim of this study is to investigate predictors of successful AF ablation in the following areas: (a) clinical factors, (b) electrophysiological, (c) electrocardiographic, (d) ultrasound, (e) cardiac anatomy, (f) biomarkers.

DETAILED DESCRIPTION:
AF is a multifactorial disease influenced by many possible mechanisms. This study will examine several different predictors of successful AF ablation: (a) clinical factors, (b) electrophysiological, (c) electrocardiographic, (d) ultrasound, (e) cardiac anatomy, (f) biomarkers. Analysis of these factors will help determine the optimal combination of predictors of successful ablation. This combination of prognostic factors can then be used to tailor therapeutic decisions specifically to individual patients and to improve patient selection for invasive treatment. Better patient selection and choice of ablation type can help increase success rates and avoid unnecessary procedures and their associated risks.

ELIGIBILITY:
Inclusion Criteria:

* paroxysmal or persistent AF
* first-time ablation of AF

Exclusion Criteria:

* patients unable to give informed consent
* serious health condition existing before ablation

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients undergoing first-time ablation (radiofrequency or pulsed field)
Sampling Method: Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-12-01 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Late AF recurrence | 3-12 months after ablation
  Late AF recurrence

SECONDARY OUTCOMES:
Late recurrence of AF or atrial tachycardia or atrial flutter | 3-12 months after ablation
  Late recurrence of AF or atrial tachycardia or atrial flutter
Early recurrence of AF | <3 months after ablation
  Early recurrence of AF
Early recurrence of AF or atrial tachycardia or atrial flutter | <3 months after ablation
  Early recurrence of AF or atrial tachycardia or atrial flutter
Time to AF recurrence and the impact of early recurrence on late AF recurrence | <3 and 3-12 months after ablation
  Time to AF recurrence and the impact of early recurrence on late AF recurrence
The superiority of monitoring using mobile health devices over traditional heart rhythm monitoring | 3 months after ablation
  The superiority of monitoring using mobile health devices over traditional heart rhythm monitoring
Progression or regression of AF | 3-12 months after ablation
  Progression of AF (from paroxysmal to persistent or persistent to permanent) or regression of AF (from persistent to paroxysmal)
Modification of treatment, including antiarrhythmic treatment | 3-12 months after ablation
  Modification of treatment, including antiarrhythmic treatment
AF-related quality of life and symptoms | Before, 3 and 12 months after ablation
  AF-related quality of life and symptoms
Periprocedural complications | Around ablation
  Periprocedural complications (e.g. cardiac tamponade, vascular complications, pseudoaneurysm, arteriovenous fistula, stroke, transient ischemic attack)
Heart rate variability and rate | <3 months after ablation
  Heart rate variability and rate
Blood biomarker levels | Before, 3 and 12 months after ablation
  Blood biomarker levels
Ablation procedure parameters | At ablation
  Ablation procedure parameters (e.g. ablation time, procedure time, number of applications, amount of painkillers used)
Cardiac remodelling | Before, 3 and 12 months after ablation
  Cardiac remodelling based on transthoracic and transesophageal echocardiography parameters

CONTACTS AND LOCATIONS:
Overall Officials: Monika Gawałko, MD, PhD, Principal Investigator — 1st Department of Cardiology, Medical University of Warsaw; Paweł Balsam, MD, PhD, Principal Investigator — 1st Department of Cardiology, Medical University of Warsaw
Locations (1):
- Medical University of Warsaw, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: Undecided